CLINICAL TRIAL: NCT00157794
Title: EnPulse Trial on Search AV+ Influence
Brief Title: EnTRINSIC - EnPulse Trial on Search AV+ Influence
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol pre-specified interim analysis showed that difference between groups was too small to reach significance.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEN_G_CA_2
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-02

CONDITIONS: Arrhythmia, Sinus
Keywords: Sinus Node Disease; Pacemaker; Dual Chamber Pacemaker
MeSH Terms: conditions — Arrhythmia, Sinus; Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Search AV+ algorithm

SUMMARY:
Right ventricular apical pacing in patients treated with a pacemaker is unnecessary in cases where patients have stable atrioventricular (AV)-conduction. Recent findings demonstrate that pacing even might have unfavourable effects, especially if patients suffer from additional cardiac diseases such as heart failure. The Search AV+ algorithm was designed to avoid ventricular pacing and support intrinsic AV-conduction in order to avoid possible detrimental effects of right ventricular apical pacing. The goal of the EnTRINSIC study is to assess the amount of ventricular stimulation, the amount of hospitalizations, the occurrence of atrial fibrillation and the usage of drugs in patients treated with pacemakers with an activated Search AV+ algorithm versus patients treated with an individual optimization of the pacemaker settings to minimize the amount of right ventricular pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sinus node disease and an intrinsic AV delay of maximal 260 ms
* Patients treated with a Medtronic pacemaker with Search AV+ algorithm

Exclusion Criteria:

* Patients with documented persistent atrial fibrillation within 6 months before implantation and slow AV-conduction
* New York Heart Association (NYHA) III/IV
* Instable angina pectoris
* Heart valve vitium
* Persistent AV-block II and III
* Early diastolic mitral regurgitation
* Implantable cardioverter defibrillator
* Participation in other clinical studies
* Pregnancy or unreliable birth control
* AV-block under strain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2004-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Amount of right ventricular pacing | Baseline to 36 months post-implant

SECONDARY OUTCOMES:
Change in intrinsic AV delay | Baseline to 36 months post-implant
Hospitalizations because of symptomatic heart failure | Baseline to 36 months post-implant
Hospitalizations because of symptomatic atrial fibrillation | Baseline to 36 months post-implant
Medication | Baseline to 36 months post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jakob, MD, Principal Investigator — Knappschaftskrankenhaus Sulzbach; Peter Lamm, MD, Principal Investigator — Klinikum der Universität München Großhadern
Locations (14):
- Germany (14):
  - Klinikum Großhadern Herzchirurgische Klinik und Poliklinik, Munich, Bavaria
  - Internistische Praxis Dr. Med. Schade, Berlin
  - St. Josefs Hospital, Bochum
  - Praxis Dr. Med. Markert, Gaggenau
  - Krankenhaus Martha Maria Halle, Halle
  - Universitätsklinikum Heidelberg, Heidelberg
  - St. Vincentius Kliniken, Karlsruhe
  - Vinzentius Krankenhaus, Landau
  - Klinikum der Johannes-Gutenberg-Universität, Mainz
  - Städtisches Klinikum Neunkirchen, Neunkirchen
  - Kreiskrankenhaus Ottweiler, Ottweiler
  - Knappschaftskrankenhaus Sulzbach, Medizinische Klinik, Sulzbach
  - Josephs-Hospital, Warendorf
  - Gemeinschaftspraxis Dr. Tamm/Dr. Hon, Wittenberg

REFERENCES:
- See also: Knappschaftskrankenhaus Sulzbach — http://www.kk-sulzbach.de
- See also: Klinikum der Universität München -Großhadern — http://hch.klinikum.uni-muenchen.de